CLINICAL TRIAL: NCT04922593
Title: A Study to Evaluate the PK Profiles of LY03010 and Relative Bioavailability at Steady-state of LY03010 Versus INVEGA SUSTENNA in Schizophrenia Patients
Brief Title: Relative Bioavailability of LY03010 Compared to Listed Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03010/CT-USA-103
Record Dates: First submitted 2021-04-27; First posted 2021-06-10 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia; Psychotic Disorders; Mood Disorders; Schizophrenia Spectrum; Mental Disorders; Antipsychotic Agents; Tranquilizing Agents; Central Nervous System Depressants; Physiological Effects of Drugs; Psychotropic Drugs; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action
Keywords: Schizophrenia; Paliperidone Palmitate; Serotonin 5-HT2 Receptor Antagonists; Serotonin Antagonists; Serotonin Agents; Dopamine D2 Receptor Antagonists; Dopamine Antagonists; Dopamine Agents
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mood Disorders; Mental Disorders | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY03010 treatment group (Experimental): LY03010 (paliperidone palmitate) is a pharmaceutical equivalent drug product to the listed drug (LD) product INVEGA SUSTENNA. The chemical name is (±)-3-[2-[4-(6-fluoro-1,2-benzisoxazol-3yl)piperidinyl]ethyl]-6,7,8,9-tetrahydro-2-methyl-4oxo-4Hpyrido[1,2-a]pyrimidin-9-yl hexadecanoate. Its molecular formula is C39H57FN4O4 and its molecular weight is 664.89 g/mol.
  LY03010 is white to off-white sterile aqueous extended-release suspension of paliperidone palmitate for IM injection. In LY03010 treatment group, all subjects will receive the first dose of 351 mg IM injection on Day 1 in the deltoid muscle, followed by five (5) monthly dosing of 156 mg IM injection in the gluteal muscle with the last dose on Day 141.
  Interventions: Drug: LY03010; paliperidone palmitate
- INVEGA SUSTENNA treatment group (Active Comparator): INVEGA SUSTENNA (234 mg, 156 mg) is manufactured by Janssen Pharmaceuticals, Inc and is commercially available. INVEGA SUSTENNA is provided in a prefilled syringe (cyclic-olefin-copolymer) with a plunger stopper and tip cap (bromobutyl rubber).
  In SUSTENNA treatment group, all subjects will receive the first dose of 234 mg IM injection in the deltoid muscle on Day 1, and a second dose of 156 mg of IM injection in the deltoid muscle on Day 8, followed by five (5) monthly dosing of 156 mg IM injection in the gluteal muscle with the last dose on Day 148.
  Interventions: Drug: INVEGA SUSTENNA

INTERVENTIONS:
Drug: LY03010; paliperidone palmitate — LY03010 is white to off-white sterile aqueous extended-release suspension of paliperidone palmitate for IM injection.
  Arms: LY03010 treatment group
Drug: INVEGA SUSTENNA — INVEGA SUSTENNA (234 mg, 156 mg) is manufactured by Janssen Pharmaceuticals, Inc and is commercially available.
  Arms: INVEGA SUSTENNA treatment group

SUMMARY:
This is a randomized, multiple-dose, open-label, parallel-group study. Subjects will undergo screening evaluations to determine eligibility within 28 days prior to study drug administration. Approximately 280 eligible subjects will be randomized in a 1:1 ratio into 1 of 2 treatment groups. Subjects will be admitted to the clinical facilities the day before dosing (Day 0), and will be randomized and receive the first dosing on Day 1. Subjects will stay at site till Day 2 after PK collection. All subjects will return to the clinical sites at designated study days for dosing, PK sample collections and assigned clinical activities.

All subjects randomized to LY03010 treatment group will receive the first dose of 351 mg LY03010 by IM injection on Day 1 in the deltoid muscle, followed by five (5) monthly dosing of 156 mg LY03010 in the gluteal muscle with the last dose on Day 141. All subjects randomized to SUSTENNA treatment group will receive the first dose of 234 mg SUSTENNA by IM injection on Day 1 in the deltoid muscle, and a second IM dose of 156 mg SUSTENNA on Day 8 in the deltoid muscle, followed by five (5) monthly IM dosing of 156 mg of SUSTENNA in the gluteal muscle with the last dose on Day 148.

End of Study (EOS) visit for LY03010 treatment group will be on Day 169, 28 days after last dosing day; End of Study for SUSTENNA treatment group will be on Day 176, 28 days after last dosing. At EOS visit, subjects will complete the study after a series of assigned clinical assessments. A 30-day follow up call will be conducted by the clinical research staff to ensure participant's well-being.

DETAILED DESCRIPTION:
This is a randomized, multiple-dose, open-label, parallel-group study. Subjects will undergo screening evaluations to determine eligibility within 28 days prior to study drug administration. Approximately 280 eligible subjects will be randomized in a 1:1 ratio into 1 of 2 treatment groups. Subjects will be admitted to the clinical facilities the day before dosing (Day 0), and will be randomized and receive the first dosing on Day 1. Subjects will stay at site till Day 2 after PK collection. All subjects will return to the clinical sites at designated study days for dosing, PK sample collections and assigned clinical activities.

All subjects randomized to LY03010 treatment group will receive the first dose of 351 mg LY03010 by IM injection on Day 1 in the deltoid muscle, followed by five (5) monthly dosing of 156 mg LY03010 in the gluteal muscle with the last dose on Day 141. All subjects randomized to SUSTENNA treatment group will receive the first dose of 234 mg SUSTENNA by IM injection on Day 1 in the deltoid muscle, and a second IM dose of 156 mg SUSTENNA on Day 8 in the deltoid muscle, followed by five (5) monthly IM dosing of 156 mg of SUSTENNA in the gluteal muscle with the last dose on Day 148.

On the day before the last dosing day visit (Day 140 for LY03010 treatment group and Day 147 for SUSTENNA treatment group), subjects will come to the clinical facility and stay at sites for 8 days for PK collection and other assigned activities. The schedules of assessments for each treatment group are listed in Table 2 and Table 3.

End of Study (EOS) visit for LY03010 treatment group will be on Day 169, 28 days after last dosing day; End of Study for SUSTENNA treatment group will be on Day 176, 28 days after last dosing. At EOS visit, subjects will complete the study after a series of assigned clinical assessments. A 30-day follow up call will be conducted by the clinical research staff to ensure participant's well-being.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, patients must meet all inclusion criteria at screening:

1. Capable of giving informed consent and complying with study procedures.
2. Have an identified support person (e.g., family member, case worker, social worker) who is considered reliable by the Investigator to help ensure compliance with study visits and to alert staff of any issues of concern.
3. Have a stable place of residence for the 3 months prior to screening and throughout the study.
4. Male or female ≥18 to ≤65 years of age who meets diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) for at least 1 year before screening.
5. Be on a stable dose of oral antipsychotic medication(s) other than risperidone, paliperidone, clozapine, ziprasidone, or thioridazine for at least 4 weeks prior to screening.
6. Be clinically stable based on clinical assessments and a Positive and Negative Syndrome Scale (PANSS) total score ≤75 as well as a PANSS HATE (hostility, anxiety, tension and excitement) subtotal score <16 at screening.
7. Clinical Global Impression-Severity (CGI-S) score of 1 to 4, inclusive.
8. For patients with schizoaffective disorder only: Young Mania Rating Scale (YMRS) ≤12 and Hamilton Rating Scale for Depression, 21-item version (HAM-D-21) ≤12.
9. Body mass index (BMI) ≥17.0 and ≤ 37 kg/m2; body weight ≥ 50 kg.
10. All female patients (childbearing potential and non-childbearing potential) must have a negative pregnancy test result at both screening and baseline. Female patients must meet 1 of the following 3 conditions: (i) postmenopausal for at least 12 months without an alternative medical cause, (ii) surgically sterile (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal occlusion) based on patient report, or (iii) if of childbearing potential (WOCBP) and heterosexually active, practicing or agree to practice a highly effective contraception method of birth control. Highly effective methods of birth control include an intrauterine device (IUD), intrauterine hormone-releasing system (IUS), and contraceptives (oral, skin patches, or implanted or injectable products) using combined or progestogen-only hormonal contraception associated with inhibition of ovulation. A vasectomized male partner is an acceptable birth control method if the vasectomized partner is the sole sexual partner of the female patient and the vasectomized partner has received medical confirmation of surgical success. Highly effective methods of birth control must be used for at least 14 days prior to study drug dosing, throughout the study, and for at least 200 days after the end-of-study (EOS) visit to minimize the risk of pregnancy.
11. Sexually active fertile male patients must be willing to use acceptable contraception methods (such as double barrier methods of a combination of male condom with either cap, diaphragm or sponge with spermicide) from study drug dosing, throughout the study, and for at least 200 days after the EOS visit if their partners are women of childbearing potential.

Exclusion Criteria:

Patients will be excluded from study entry if 1 or more exclusion criteria are met at screening:

1. Primary and active DSM-V Axis I diagnosis other than schizophrenia or schizoaffective disorder.
2. Patients who meet DSM-V criteria for substance abuse (moderate or severe), or test positive for a drug of abuse or alcohol at screening or baseline with the exception of 1) caffeine or nicotine in the past 6 months prior to screening, or 2) test positive for barbiturate or benzodiazepine which can be accounted for by documented prescriptions from a treating physician as a part of the treatment for the patient's psychiatric illness.
3. Patients who received any of following treatment:

   * Use of oral risperidone or paliperidone within 2 weeks before screening.
   * Use of Clozapine, Thioridazine or Ziprasidone within 4 weeks before screening.
   * Use of 2-week depot formulation of risperidone (RISPERDAL CONSTA) within 3 months, 1-month depot formulation of risperidone (PERSERIS KIT) or 9-hydroxy risperidone (INVEGA SUSTENNA) within 1 year, or 3-month depot formulation of 9-hydroxy risperidone (INVEGA TRINZA) within 2 years before screening. Use of other long-acting injectable for the treatment of schizophrenia within 4 weeks before screening.
   * Use of nonselective or irreversible monoamine oxidase inhibitor (MAOI) antidepressants within 30 days before screening. Patients on other antidepressants should be excluded as well unless the dose has been stable for more than 30 days before screening.
   * Use of strong inducers or inhibitors of CYP3A4 or P-glycoprotein (P-gp) within 2 weeks or 5 half lives, whichever is longer, before screening.
   * Electroconvulsive therapy within 60 days before screening.
4. Known or suspected hypersensitivity or intolerance of risperidone, paliperidone, or any of their excipients (oral risperidone tolerability test will be completed during the screening period, approximately14 days but no less than 9 days prior to dosing, for patients without documented evidence [medical record or written statement from a licensed medical practitioner who has treated the patient] of tolerating risperidone or paliperidone, and patients who show an allergic reaction to this test will be excluded from the study).
5. Patients who pose a significant risk of a suicide attempt based on history or the Investigator's judgment; answer "yes" to Suicidal Ideation items 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) for current or past 6 months on the "Baseline/Screening version" at screening; have had suicidal behavior in the last 6 months as measured by the C-SSRS at screening; or are at imminent risk of suicide or violent behavior based on the Investigator's clinical assessment or the C-SSRS assessment of lifetime suicidal ideation or behavior at screening.
6. Any one or more of the following 3 conditions: (i) clinically significant liver dysfunction, (ii) hepatitis B surface antigen (HBsAg) positive, hepatitis C (HCV) positive, or (iii) a serum alanine transaminase (ALT) or aspartate transaminase (AST) > 2x upper limit of normal (ULN) range; or a total bilirubin > 1.5 x ULN(if the ALT or AST levels are between 2x and 3x ULN in the first screening test and the elevation may be caused by non-specific reasons in the judgment of the Investigator, a second test can be performed after one week. If the repeated ALT or AST levels are still >2x ULN, the patient must be excluded from the study. Patients who are HCV antibody reactive but confirmed HCV RNA not detected may be enrolled, if this condition has been previously considered stable without treatment or after the completion of appropriate treatment, and liver function is normal.
7. History of symptomatic orthostatic hypotension or with a decrease of ≥ 20 mmHg in systolic blood pressure (SBP) or decrease of ≥10 mmHg in diastolic blood pressure (DBP) when changing from supine to standing position after having been in the supine position for at least 5 minutes or SBP less than 105 mmHg in a supine position prior to randomization.
8. Uncontrolled diabetes or hemoglobin A1c (HbAlc) level ≥ 7% at screening.
9. Indication of impaired renal function at Screening (estimated glomerular filtration rate < 80 mL/min).
10. History of neuroleptic malignant syndrome (NMS) or tardive dyskinesia; history of severe akathisia or extra-pyramidal reactions such as dystonia with previous use of risperidone or other neuroleptic treatments; score ≥ 3 on the Global Clinical Assessment of the BARS or score ≥ 2 on the AIMS at screening.
11. QTcF interval greater than 450 msec for males and 460 msec for females at screening, or other clinically significant ECG findings in the opinion of the Investigator.
12. Clinically significant past medical history (within 2 years) of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, renal, hepatic, bronchopulmonary, neurologic, immunologic disorders, or drug hypersensitivity which, in the judgment of the Investigator, would interfere with the patient's ability to participate in the study.
13. Subject has clinical signs and symptoms consistent with Coronavirus disease 2019 (COVID-19), e.g., fever, dry cough, dyspnea, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 30 days prior to screening or on admission.
14. Subject who had severe course of COVID-19 (i.e., hospitalization, extracorporeal membrane oxygenation (ECMO), and/or mechanically ventilated).
15. Malignancies within 5 years with the exception of cured basal cell or squamous cell skin cancer or in situ cervical cancer prior to screening.
16. History or current diagnosis of epilepsy or convulsive disorder other than a single childhood febrile seizure.
17. History or current diagnosis of Parkinson's diseases, Dementia with Lewy Bodies or other Dementia-related psychosis.
18. Receipt of another investigational product within 1 month, or 5 half-lives of the other investigational product, whichever is longer, prior to screening.
19. Donation or blood collection of > 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening.
20. Clinical Laboratory at screening indicating white blood cells <3x109/L, or neutrophils <1.5x109/L or platelets < 80 x109/L.
21. Has a prolactin laboratory value ≥ 100 ng/ml at screening.
22. Human immunodeficiency virus (HIV) test positive.
23. Any clinical observation or clinical laboratory abnormality findings at screening or baseline visits which, in the opinion of the Investigator, may endanger the patient or interfere with the endpoints of the study. If the results of clinical laboratory testing are outside normal reference ranges, the patient may be enrolled but only if these findings are determined not to be clinically significant by the Investigator. This determination must be recorded in the patient's source documents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
The relative bioavailability of LY03010 versus INVEGA SUSTENNA at steady-state | 176 days
  The relative bioavailability of LY03010 versus INVEGA SUSTENNA will be evaluated by the analysis of the area under the plasma concentration-time curve over a dosing interval at steady state (AUCtau-ss) of plasma paliperidone.
Relative Bioavailability of LY03010 compared to Listed Drug | 176 days
  The relative bioavailability of LY03010 versus INVEGA SUSTENNA will be evaluated by the analysis of maximum peak steady-state (Cmax-ss) of plasma paliperidone concentration during a dosage interval.

SECONDARY OUTCOMES:
Compare the PK profile between LY03010 and INVEGA SUSTENNA at the initial phase | 36 days
  AUC of paliperidone from the two different initial dosing regimens will be compared.
Compare the PK profile between the two treatments at the initial phase. | 36 days
  Cmax of paliperidone from the two different initial dosing regimens will be compared.
Compare the PK profile between the two treatments. | 36 days
  Cmin of paliperidone from the two different initial dosing regimens will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Li, MD, Study Chair — Luye Pharma US Ltd
Locations (9):
- United States (9):
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - CNS Network, LLC, Torrance, California
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - Uptown Research Institute, LLC, Chicago, Illinois
  - Hassman Research Institute, Berlin, New Jersey
  - Hassman Research Institute, Marlton, New Jersey
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No